CLINICAL TRIAL: NCT04524221
Title: A Phase 1b Study of PTG-100 in Patients With Celiac Disease
Brief Title: PTG-100 for Patients With Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nielsen Fernandez-Becker (Other)
Collaborators: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nielsen Fernandez-Becker, Clinical Associate Professor, Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 57613; PTG-100-05-CeD (Other: Stanford University)
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — PTG-100 peptide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTG-100 (Experimental): Patients will receive either placebo (fake drug) or PTG-100 (real drug) in capsule form twice daily for 42 days.
  Interventions: Drug: PTG-100
- Placebo (Placebo Comparator): Patients will receive either placebo (fake drug) or PTG-100 (real drug) in capsule form twice daily for 42 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTG-100 — PTG-100, 600mg taken twice daily in capsule form for 42 days
  Arms: PTG-100
Drug: Placebo — Placebo taken twice daily in capsule form for 42 days
  Arms: Placebo

SUMMARY:
The goal of this study is to learn whether or not the drug PTG-100 can reduce or prevent inflammatory injury to the small intestine that occurs when people with celiac disease eat food products containing gluten.

This is a clinical research study to determine the safety and efficacy of PTG-100 in preventing gluten-induced inflammatory injury to the small intestine in patients with celiac disease. 30 patients will receive either placebo (fake drug) or PTG-100 (real drug) in capsule form twice daily for 42 days. They will also receive a gluten challenge twice daily in the form of a cookie or equivalent. An upper gastrointestinal endoscopy and exam including small bowel mucosa biopsy will be performed at the start of the treatment period and again at the end. Blood samples will be routinely taken to evaluate safety and the drug's mechanism of action throughout the study, and symptoms will be recorded using the celiac symptoms index (CSI) survey.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of celiac disease

Exclusion Criteria:

* Active GI disease or history of clinically significant diseases
* Diagnosis of Crohn's disease or ulcerative colitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Percentage change in villous height-to crypt ratio | 42 days
  Percentage change from baseline to Week 6 in villous height-to crypt depth (Vh:Cd) ratio

SECONDARY OUTCOMES:
Change in celiac disease antibodies | 42 days
  Changes in anti-tTG antibodies from baseline
Changes in celiac disease antibodies | 42 days
  Changes in anti-DGP antibodies from baseline
CD3- positive intraepithelial lymphocyte density | 42 days
  CD3- positive intraepithelial lymphocyte density
Celiac symptom index (CSI) | 42 days
  Changes in validated celiac symptom index (CSI)
Characterization of immune modulators underlying mechanism of action in celiac disease. | 42 days
  Identification of immune cell populations targeted by PTG-100 to better understand mechanism of action in celiac disease in both blood and tissue temporally following exposure to drug.

CONTACTS AND LOCATIONS:
Overall Officials: Nielsen Q Fernandez-Becker, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No